CLINICAL TRIAL: NCT06531187
Title: Applying Innovative Gamification Education in Evidence-Based Practice for Clinical Nurses
Brief Title: Gamification Design in Evidence-Based Education for Clinical Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ling-Yu Chien (Other)
Responsible Party: Sponsor-Investigator, Ling-Yu Chien, Researcher, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B202005016
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Nursing Education; Evidence-Based Practice
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gamified group (Experimental): The experimental group will receive a 4-hour gamified instructional design course focused on teaching Evidence-Based Practice (EBP), based on the Octalysis Framework of game elements proposed by Chou (2019).
  Interventions: Other: Evidence-Based Practice (EBP) Teaching
- conventional small group discussion (Active Comparator): The active comparator group will participate in 4-hour conventional small group discussions focused on teaching Evidence-Based Practice (EBP).
  Interventions: Other: Evidence-Based Practice (EBP) Teaching

INTERVENTIONS:
Other: Evidence-Based Practice (EBP) Teaching — The experimental group will receive a 4-hour gamified instructional design course focused on teaching Evidence-Based Practice (EBP), based on the Octalysis Framework of game elements proposed by Chou (2019).
  The active comparator group will participate in 4-hour conventional small group discussions focused on teaching Evidence-Based Practice (EBP).

SUMMARY:
The goal of this study is to compare the effectiveness of gamification versus group discussion in evidence-based practice (EBP) education for clinical nurses. It aims to improve learning outcomes and clinical application of EBP.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

Does gamification enhance the knowledge acquisition of clinical nurses in EBP? What barriers to evidence-based practice do nurses face? How does gamification affect cognitive load, self-efficacy, and attitudes towards EBP? Researchers will compare gamification to traditional group discussion methods to evaluate their impact on clinical practice.

Participants will:

Be clinical nurses from Tri-Service General Hospital with varying ranks and experiences.

Be randomly assigned to either the gamification group or the control group. Participate in EBP courses based on their clinical rank and experience. Complete pre- and post-intervention assessments and a six-month follow-up. Data collection will measure barriers to evidence-based practice, cognitive load, knowledge acquisition, self-efficacy, attitudes, course satisfaction, and practical application through written reports. Data analysis will use descriptive and inferential statistics to evaluate the effectiveness of the interventions.

This study aims to provide evidence on the most effective teaching methods for EBP, contributing to improved educational strategies and better clinical practices for nurses.

ELIGIBILITY:
Inclusion Criteria:

* Active clinical nurses aged 20-65. Clinical nurses within the hospital who registered for the workshop via e-learning.

Nurses with more than three months of work experience and a signed contract.

Exclusion Criteria:

* Nurses with less than three months of work experience or without a signed contract.

Participants cannot simultaneously attend both types of courses. Nurses at level N2 or above, nurses from other hospitals, nurse practitioners, or nursing supervisors are not included in this study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
EBP Competence | Baseline, immediately after the workshop, and 6 months follow-up
  Measured using the ACE tool developed by Ilic et al. (2014).
Self-Efficacy and attitudes | Baseline, immediately after the workshop, and 6 months follow-up
  Assessed using the Taipei Evidence-Based Practice Questionnaire (TEBPQ) (Chen et al., 2014).
Participant Satisfaction with EBP Teaching | immediately after the workshop
  Measured using a questionnaire designed specifically for this study.
practicing applicability | 6 months follow-up
  The patient care report was then submitted for a panel of experts' review.

SECONDARY OUTCOMES:
Cognitive Load | Baseline, and 6 months follow-up
  Assessed using items referenced from Albarqouni et al. (2018).
Barriers | Baseline, and 6 months follow-up
  Measured using the Chinese Evidence-Based Practice Scales (Wang et al., 2012).

CONTACTS AND LOCATIONS:
Overall Officials: Ling-Yu Chien, Study Director — National Defense Medical Center, Taiwan
Locations (1):
- National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No